CLINICAL TRIAL: NCT06970639
Title: A Phase III, International, Multicenter, Randomized, Controlled, Open-label Clinical Study Evaluating Furmonertinib Plus Platinum-based Doublet Chemotherapy Versus Osimertinib in Patients With Epidermal Growth Factor Receptor (EGFR) Sensitizing Mutation-Positive Non-squamous Non-Small Cell Lung Cancer (NSCLC) and Brain Metastases
Brief Title: A Study Evaluating Furmonertinib Plus Platinum-based Doublet Chemotherapy Versus Osimertinib in Patients With Epidermal Growth Factor Receptor (EGFR) Sensitizing Mutation-Positive Non-squamous Non-Small Cell Lung Cancer (NSCLC) and Brain Metastases
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Allist Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALSC014AST2818
Record Dates: First submitted 2025-04-09; First posted 2025-05-14 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-03

CONDITIONS: NSCLC Patients With Brain Metastasis
Keywords: EGFR; firmonertinib
MeSH Terms: interventions — Carboplatin; Cisplatin; Injections; Pemetrexed; osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Furmonertinib combined with chemotherapy (Experimental): Furmonertinib Mesilate Tablets+Carboplatin Injection/Cisplatin for injection+Pemetrexed Disodium for Injection
  Interventions: Drug: Furmonertinib Mesilate Tablets; Drug: Carboplatin Injection; Drug: Cisplatin for injection; Drug: Pemetrexed Disodium for Injection
- Osimertinib Mesylate Tablets (Active Comparator): Osimertinib Mesylate Tablets
  Interventions: Drug: Osimertinib Mesylate Tablets

INTERVENTIONS:
Drug: Furmonertinib Mesilate Tablets — Usage and dosage: 80mg, 240mg, or 160mg QD orally Medication duration: A cycle of 21 days until intolerable toxicity, disease progression, death, or initiation of new anti-tumor therapy occurs
  Arms: Furmonertinib combined with chemotherapy
Drug: Carboplatin Injection — Usage and dosage: Administer via IV infusion, with a dosage of AUC5, not exceeding 750 mg.
  Medication schedule: every 3 weeks as a cycle, D1 administration per cycle, immediate administration of carboplatin upon completion of pemetrexed infusion, intravenous infusion, carboplatin can be used for up to 4 cycles.
  Arms: Furmonertinib combined with chemotherapy
Drug: Cisplatin for injection — Usage and dosage: Administer via IV infusion at a dose of 75 mg/m2. Medication schedule: Every 3 weeks as a cycle, with D1 administration per cycle. Cisplatin is administered approximately 30 minutes after the infusion of pemetrexed, via intravenous infusion. Adequate hydration therapy must be received before and after cisplatin treatment. Cisplatin can be used for up to 4 cycles.
  Arms: Furmonertinib combined with chemotherapy
Drug: Pemetrexed Disodium for Injection — Usage and dosage: Intravenous (IV) infusion administration, dosage of 500 mg/m2 Medication schedule: Administer on the first day of each cycle (21 days per cycle, i.e. every 3 weeks) until intolerable toxicity, disease progression, death, or initiation of new anti-tumor therapy occurs.
  Arms: Furmonertinib combined with chemotherapy
Drug: Osimertinib Mesylate Tablets — Usage and dosage: 80mg, QD administration Medication duration: A cycle of 21 days until intolerable toxicity, disease progression, death, or initiation of new anti-tumor therapy occurs
  Arms: Osimertinib Mesylate Tablets

SUMMARY:
This study is a Phase III, international, multicenter, randomized, controlled, open-label clinical trial. The primary objective is to evaluate the efficacy and safety of furmonertinib plus platinum-based doublet chemotherapy (Arm A) versus osimertinib monotherapy (Arm B) in patients with EGFR sensitizing mutation-positive non-squamous non-small cell lung cancer (NSCLC) and brain metastases. Additionally, a proportion of subjects will receive furmonertinib monotherapy (Arm C) to further explore its efficacy and safety profile.

Stage 1 is the safety run-in phase, planned to enroll approximately 30 subjects who will be randomized at a 1:1 ratio to receive either furmonertinib 80 mg QD plus platinum-based chemotherapy or furmonertinib 160 mg QD plus platinum-based chemotherapy, aiming to evaluate the safety and tolerability of different furmonertinib doses in combination with platinum-based chemotherapy.

Stage 2 is the randomized controlled phase, in which approximately 350 subjects will be randomized in a 3:3:1 ratio (Arm A : Arm B : Arm C) to receive the investigational treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the trial and voluntarily sign the informed consent form;
2. Age ≥18 years at the time of signing ICF, regardless of gender;
3. Histologically/cytologically confirmed non-squamous NSCLC with brain parenchymal metastases assessed by BICR; Subjects with both brain parenchymal and leptomeningeal metastases are eligible. Subjects without brain metastases may be enrolled in the safety run-in phase.
4. For subjects with brain metastases: clinically stable for ≥4 weeks prior to first dose AND no requirement for corticosteroids/anticonvulsants for ≥14 days prior to first dose; Investigator-confirmed no need for local therapy for brain metastases during screening.
5. Confirmed EGFR sensitizing mutations (ex19del or L858R) via tumor tissue/cytology/blood testing;
6. No prior systemic anti-tumor therapy for advanced/metastatic NSCLC; Subjects who received (neo)adjuvant chemotherapy or definitive chemoradiotherapy must have disease recurrence/progression ≥6 months after completion;
7. ≥1 measurable intracranial AND extracranial lesion(s) per RECIST v1.1 without prior local treatment;
8. ECOG PS 0-1 with no deterioration within 2 weeks prior to first dose, and life expectancy ≥3 months;
9. Adequate bone marrow and organ function (no transfusion/G-CSF within 2 weeks prior to first dose);
10. All prior treatment-related toxicities resolved to ≤Grade 1 (per NCI CTCAE v5.0) except alopecia (≤Grade 2) or peripheral neuropathy (≤Grade 2);
11. Women of childbearing potential (WOCBP) must have negative serum pregnancy test within 7 days prior to first dose, be non-lactating, and use effective contraception from ICF signing until 6 months after last dose. Male subjects with fertile partners must use contraception during the same period.

Exclusion Criteria:

1. The tumor histology or cytology confirmed that the combination of neuroendocrine carcinoma, sarcomatoid carcinoma or squamous cell carcinoma was more than 10%;
2. Known subjects with ALK positive, ros1 positive, RET fusion positive, ntrk fusion positive, BRAF V600 mutation, met exon 14 skipping variant and other approved drugs for this target;
3. Subjects with meningeal metastasis but no brain parenchymal metastasis confirmed by MRI and / or CSF malignant cell examination;
4. Subjects who have previously received any of the following treatments:

   1. Have received any systemic anti-tumor therapy targeting EGFR in the past, including those in clinical research stage (including EGFR TKI, monoclonal antibody, bispecific antibody, etc.);
   2. Previously received systemic antitumor therapy (such as chemotherapy, targeted therapy, immunotherapy, etc.) for locally advanced / metastatic non-small cell lung cancer;
   3. Received > 30 Gy of chest radiotherapy within 6 months before the first dose; Received non thoracic radiotherapy of >30 Gy within 4 weeks before the first dose; Received palliative radiotherapy ≤ 30Gy within 2 weeks before the first dose; Previous brain radiotherapy;
5. Chinese patent medicine that has received non-specific immune modulators (including but not limited to interferon and IL-2) and approved anti-tumor indications within 2 weeks before the first administration;
6. Have used any strong inhibitor of cytochrome P450 3A4 (CYP3A4) within 7 days before the first administration or any strong inducer of CYP3A4 within 21 days before the first administration;
7. Other malignant tumors in addition to the primary tumor; Skin basal cell or squamous cell carcinoma, superficial bladder cancer, cervical carcinoma in situ, breast ductal carcinoma in situ and papillary thyroid cancer that can be treated locally and have been cured can be selected; Subjects with a history of other malignancies and who have been cured for ≥ 3 years after radical treatment can be enrolled;
8. Brain metastasis subjects with known brain stem metastasis, spinal cord metastasis and / or compression; Subjects with acute or progressive intracranial hypertension related symptoms during the screening period; Subjects with brain herniation or near brain herniation; Brain imaging revealed significant brain midline deviation and other subjects requiring urgent local treatment;
9. According to CTCAE 5.0, there were subjects with grade 2 headache, vomiting, papilledema, etc. caused by increased intracranial pressure during the screening period; Subjects with grade 2 sensory / motor impairment and visual field damage caused by brain metastasis during the screening period; Subjects with mental symptoms (such as dementia, sluggish reaction, etc.) or seizures caused by brain metastasis during the screening period; Subjects who can control relevant central nervous system symptoms ≤ 1 grade by steroid hormones or anticonvulsants can be enrolled;
10. The tumor invades the surrounding important organs and blood vessels (such as the heart, esophagus, superior vena cava, etc.) or has the risk of esophago tracheal fistula or esophago pleural fistula;
11. Cardiovascular and cerebrovascular disease or cardiovascular and cerebrovascular risk factors exist.
12. There are uncontrollable systemic diseases.
13. There is a history of (non infectious) interstitial lung disease (ILD) or non infectious pneumonia requiring steroid treatment.
14. Pulmonary complications lead to clinically severe lung damage.
15. Severe acute or chronic infection
16. Subjects who are receiving long-term systemic corticosteroid therapy with prednisone > 10 mg/d or equivalent anti-inflammatory active drugs or any form of immunosuppressive therapy before the first administration [subjects who need bronchodilators, inhaled or topical steroids or local steroid injection therapy, or as preventive medication for hypersensitivity reactions (such as medication before CT examination, etc.), or to control central nervous system symptoms in patients with brain metastasis can be included in the study];
17. Subjects who had undergone major surgery within 4 weeks before the first dose or were expected to undergo major surgery during the study;
18. Bleeding symptoms with significant clinical significance or obvious bleeding tendency within 4 weeks before the first administration.
19. Severe gastrointestinal dysfunction is known.
20. Known or suspected allergy to the ingredients of the study drug or its analogues;
21. Pregnant or lactating women or female subjects who plan to become pregnant during the study or within 6 months after the last dose;
22. In the judgment of the investigator, the subject has other factors that may affect the results of the study or cause the forced termination of the study, such as alcohol abuse, drug abuse, suffering from other serious diseases (including mental diseases) requiring combined treatment, serious abnormal laboratory test values, family or social factors and other conditions that may affect the safety of the subject or the collection of test data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AE) | Up to 4 years
  Safe import period
Serious Adverse Event (SAE) | Up to 4 years
  Safe import period
Progression-free survival (PFS) | Up to 4 years
  Randomized Controlled Phase：PFS assessed by BICR based on recist1.1; PFS was defined as the time from the date of randomization to the date of first documented disease progression (assessed according to RECIST v1.1 criteria) or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Progression free survival (PFS) evaluated by researchers based on RECIST 1.1 | Up to 4 years
  Both the safe introduction period and randomized controlled trials require evaluation of progression free survival (PFS)
Objective response rate (ORR) | Up to 4 years
  Both the safe introduction period and randomized controlled trials require evaluation of objective response rate (ORR)
Disease control rate (DCR) | Up to 4 years
  Both the safe introduction period and randomized controlled trials require evaluation of disease control rate (DCR)
Duration of Relief (DOR) | Up to 4 years
  Both the safe introduction period and randomized controlled trials require evaluation of Duration of Relief (DOR)
Overall survival (OS) | Up to 4 years
  safe introduction period
InterPlanetary File System（iPFS） by researchers and BICR based on RECIST 1.1 evaluation | Up to 4 years
  Randomized Controlled Phase
Depth of Response（DepOR） by researchers and BICR based on RECIST 1.1 evaluation | Up to 4 years
  Randomized Controlled Phase
adverse events (AE) | Up to 4 years
  Randomized Controlled Phase
serious adverse events (SAE) | Up to 4 years
  Randomized Controlled Phase
Patient Reported Outcomes by EORTC QLQ LC13 questionnaire | Up to 4 years
  Randomized Controlled Phase：To assess the impact of firmonertinib on patients' disease-related symptoms and health related quality of life (HRQoL).
Patient Reported Outcomes by EORTCQLQ-C30 questionnaire | Up to 4 years
  Randomized Controlled Phase：To assess the impact of firmonertinib on patients' disease-related symptoms and health related quality of life (HRQoL).
Peak Plasma Concentration (Cmax) | Up to 4 years
  Randomized Controlled Phase
Steady-state oral clearance（CLss/F） | Up to 4 years
  Randomized Controlled Phase
Steady-state minimal concentration（Cmin,ss） | Up to 4 years
  Randomized Controlled Phase
Steady-state area under the curve（AUCss） | Up to 4 years
  Randomized Controlled Phase

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangdong, Guangzhou, China